CLINICAL TRIAL: NCT00643292
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin SR Versus Amoxicillin/Clavulanate Potassium (Augmentin ES-600 Trademark) for the Treatment of Acute Otitis Media in Children Undergoing Diagnostic Tympanocentesis
Brief Title: A Single, High-Dose Azithromycin Extended Release (60 mg/kg) Compared With 10 Days of High-Dose Amoxicillin Clavulanate in Children With Ear Infections at High Risk of Persistent/Recurrent Ear Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661073
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: amoxicillin/clavulanate postassium (Augmentin ES-600)
- 2 (Experimental)
  Interventions: Drug: azithromycin SR

INTERVENTIONS:
Drug: amoxicillin/clavulanate postassium (Augmentin ES-600) — amoxicillin/clavulanate postassium 90/6.4 mg/kg/day, given in divided doses q12h, for 10 days
  Arms: 1
Drug: azithromycin SR — azithromycin SR 60 mg/kg x 1 dose
  Arms: 2

SUMMARY:
A phase 3 randomized, multicenter, double blind, double dummy study to assess the efficacy, safety, and compliance of a single dose of azithromycin extended release compared with a 10-day course of amoxicillin/clavulanate twice daily in children at high risk for persistent or recurrent ear infections

ELIGIBILITY:
Inclusion Criteria:

Outpatients with clinical evidence of acute otitis media who weigh at least 5 kg were included

Exclusion Criteria:

Patients with previously diagnosed disease of immune function, treatment with any systemic antibiotic within the previous 7 days, or cleft lip/palate or other anatomic abnormality predisposing to otitis media were excluded.

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 902 (Actual)
Dates: Start 2003-01; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
clinical response (cure or failure) in the Clinical Per Protocol population | Test of Cure (TOC) visit (Day 12-14)

SECONDARY OUTCOMES:
summary of baseline susceptibilities | Study endpoint
clinical response (cure or failure) in the Clinical Per Protocol population | On-Treatment (OT) visit (Day 4-6)
Laboratory abnormalities | Baseline and TOC visit
bacteriological response (eradication, presumed eradication, persistence, or presumed persistence) on a per pathogen basis for the Bacteriological Per Protocol population | TOC visit
adverse events | Continuous
clinical response (cure or failure) in all populations except the Clinical Per Protocol population | OT visit and TOC visit
clinical response (cure or failure) by baseline pathogen for the Bacteriological Per Protocol population | OT visit, TOC visit, and Long-Term Follow-up (LTFU) visit (Day 28-32)
clinical response (cure or failure) in the Clinical Per Protocol population | LTFU visit
clinical scores for the Clinical Per Protocol population | OT visit and TOC visit
persistence of middle ear fluid for the Clinical Per Protocol population | TOC visit and LTFU visit
audiologic response | LTFU visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (21):
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Bellflower, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Newhall, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Pico Rivera, California
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evanston, Illinois
  - Pfizer Investigational Site, Bardstown, Kentucky
  - Pfizer Investigational Site, Springfield, Kentucky
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Payson, Utah
  - Pfizer Investigational Site, Springville, Utah
  - Pfizer Investigational Site, Vienna, Virginia
- Pfizer Investigational Site, Buenos Aires, Argentina
- Chile (3):
  - Pfizer Investigational Site, Independencia, Santiago Metropolitan
  - Pfizer Investigational Site, Recoleta, Santiago Metropolitan
  - Pfizer Investigational Site, Santiago
- Pfizer Investigational Site, San José, Provincia de San José, Costa Rica
- Pfizer Investigational Site, Santo Domingo, DN, Dominican Republic
- Estonia (4):
  - Pfizer Investigational Site, Pärsti Vald, Viljandimaa
  - Pfizer Investigational Site, Rakvere
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Pfizer Investigational Site, Guatemala City, Departamento de Guatemala, Guatemala
- Israel (4):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Litwinsky
- Pfizer Investigational Site, Chihuahua City, Chihuahua, Mexico
- Pfizer Investigational Site, Panama City, Panama
- Poland (2):
  - Pfizer Investigational Site, Chorzów
  - Pfizer Investigational Site, Lublin
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Smolensk
- Slovakia (2):
  - Pfizer Investigational Site, Košice, Slovakia
  - Pfizer Investigational Site, Martin, Slovakia
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661073&StudyName=A%20Single%2C%20High-Dose%20Azithromycin%20Extended%20Release%20%2860%20mg/kg%29%20Compared%20with%2010%20Days%20of%20High-Dose%20Amoxicillin%20Clavulanate%20in%20Children%20